CLINICAL TRIAL: NCT02832180
Title: The Effect of BMS-986142 on the Pharmacokinetics of a Combined Oral Contraceptive Containing Ethinyl Estradiol and Norethindrone Acetate in Healthy Female Subjects
Brief Title: The Effect of BMS-986142 on the Pharmacokinetics of a Combined Oral Contraceptive (OC) Containing Ethinyl Estradiol (EE) and Norethindrone Acetate (NET) in Healthy Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IM006-032
Record Dates: First submitted 2016-05-16; First posted 2016-07-14 (Estimated); Last update posted 2016-12-26 (Estimated); Status verified 2016-12

CONDITIONS: Arthritis
Keywords: Rheumatoid
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Daily single dose of OC containing EE and NET (Experimental): Daily single dose of OC Containing EE and NET alone.
  Interventions: Drug: OC containing EE and NET
- Daily single dose of OC in combination with BMS-986142 (Experimental): Daily single dose of OC containing EE and NET in combination with BMS-986142.
  Interventions: Drug: OC containing EE and NET; Drug: BMS-986142

INTERVENTIONS:
Drug: OC containing EE and NET
Drug: BMS-986142
  Arms: Daily single dose of OC in combination with BMS-986142

SUMMARY:
This is an open-label, 2-cycle, multiple-dose, single-sequence study in women of child-bearing potential. The primary objective is to assess the effect of BMS-986142 on the pharmacokinetics (PK) of Combined Oral Contraceptive Containing Ethinyl Estradiol and Norethindrone Acetate.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* Target population: Healthy females with no clinically significant deviations from normal in medical history, physical examinations, vital signs, electrocardiograms (ECGs), physical measurements, and clinical laboratory tests that are willing to switch to Loestrin during the study.
* Body Mass Index (BMI) between 18 to 32 kg/m2.
* Women of childbearing potential with intact ovarian function and history of regular menstrual cycles must have been on a stable regimen of combination of birth control containing ethinyl estradiol without evidence of clinically significant breakthrough bleeding or spotting for at least 2 consecutive months prior to Day -1.
* Women of childbearing potential must agree to follow instructions for method(s) of contraception for the duration of treatment with study drugs (53 days) plus 5 half-lives of BMS-986142 (3 days) plus 30 days (duration of ovulatory cycle) for a total of 86 days.

Exclusion Criteria:

* History of any chronic or acute illness including active TB in the last 3 years, recent infection, gastrointestinal disease, smoking within less than 6 months prior to dosing, alcohol abuse, inability to tolerate oral medication, or inability to be venipunctured.
* History of jaundice or irregular bleeding associated with taking oral contraceptives, frequent headaches, cerebrovascular or coronary-artery disease, retinal vascular lesions, cancer of the breast or endometrium, deep venous thrombosis, pulmonary embolism, stroke, transient ischemic attack, or phlebitis.
* Vaccination or plans for vaccination with any live vaccine 12 weeks prior to first dose of study drug, during the course of the study, or 30 days after the last dose of study drug.
* Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, electrocardiograms, or clinical laboratory determinations beyond what is consistent with the target population.
* History of allergies and adverse drug reaction to any oral contraceptive compounds or Bruton tyrosine kinase (BTK) inhibitors.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2016-05; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of EE and NET | Cycle 1 Day 21 to Cycle 2 Day 22 (30 days)
Area under the concentration-time curve (AUC) of EE and NET | Cycle 1 Day 21 to Cycle 2 Day 22 (30 days)
Area under the concentration-time curve over the dosing interval [AUC (TAU)] of EE and NET | Cycle 1 Day 21 to Cycle 2 Day 22 (30 days)

SECONDARY OUTCOMES:
Safety endpoints include the incidence of adverse events (AEs), serious adverse events (SAEs), AEs leading to discontinuation, and death. | Cycle 1 Day 1 to Cycle 2 Day 25; For SAEs up to 30 days post discontinuation of dosing or participation.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- United States (2):
  - Miami Research Associates, Miami, Florida
  - Covance Evansville Clinical Research Unit, Evansville, Indiana

REFERENCES:
- See also: BMS Clinical Trial Education Resource — http://www.bms.com/studyconnect/pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/pages/investigator_inquiry_form.aspx